CLINICAL TRIAL: NCT06565481
Title: Measurement Properties (Reliability and Validity) of a Set of Assessments Evaluating Physical Function in People with Hemophilia
Brief Title: Measurement Properties in People with Hemophilia
Acronym: HEMOPRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-01354
Record Dates: First submitted 2024-07-23; First posted 2024-08-22 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-08

CONDITIONS: Hemophilia a; Hemophilia B; Musculoskeletal Complication; Measurement Error
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — hydroxyethyl methacrylate

STUDY DESIGN:
Intervention Model Description: This study, including two time points, is performed to determine validity and reliability of performance based assessments using a one-arm sample.
  A test retest design is used to determine reliability and a cross-sectional design to determine validity.
  For each participant, the measures will be performed on two time points with a minimal recovery break of 2 days in one single centre in the Canton of Zurich (University Hospital Zurich).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Test-Re Test Arm (Other): This study, including two time points, is performed to determine validity and reliability of performance based assessments using a one-arm sample.
  A test retest design is used to determine reliability and a cross-sectional design to determine validity.
  For each participant, the measures will be performed on two time points with a minimal recovery break of 2 days in one single centre in the Canton of Zurich (University Hospital Zurich).
  Interventions: Other: Measurement Properties (Reliability and Validity) of a Set of Assessments evaluating Physical Function in adult Participants with Hemophilia

INTERVENTIONS:
Other: Measurement Properties (Reliability and Validity) of a Set of Assessments evaluating Physical Function in adult Participants with Hemophilia — This study evaluates the reliability (Test-Retest) of six health related instruments that assess physical function in people with hemophilia: Short Physical Performance Battery, Unipedal Stance Test, Four Square Step Test, Timed up and Go, 1 kg Arm Lift Test, 30 Second Chair Stand Test. This study is needed to determine the psychometric properties of these six assessments. Validity of these test will be determined with the Short Form 36, the Hemophilia Activities List and the Hemophilia Joint Health Score Methodology: Reliability (Test re-test study and validity (cross sectional study) of the six tests reported in patients with hemophilia.
  This intervention contains physiotherapie assessments, however, no drugs nor medical devices.

SUMMARY:
The aim of this project is to determine the measurement properties (namely reliability and validity) of a set of clinical assessments, measuring different aspects of physical function.

DETAILED DESCRIPTION:
The medical treatment of hemophilia has advanced greatly in recent years. There are now medications that reduce the physical symptoms of hemophilia. Nevertheless, those affected by hemophilia suffer from restricted mobility, reduced strength, reduced balance and pain as a result of the repeated bleeding. In order to make well-founded decisions regarding possible supportive therapeutic or medical measures, it is important to be able to estimate the extent of such limitations and whether these will change or remain stable.

The study is needed to validate the measurement properties of measurement instruments used to measure the effects of physical training interventions in participants with hemophilia. Clinical questions can only be solved if measuring instruments with sufficient measuring properties are used. These measurement properties must be evaluated in a relevant population. Otherwise, health professionals cannot assess whether measures or treatment are not effective or whether measured changes are not large enough to detect an actual change. Therefore, research is required to ensure that adequately studied measurement instruments are available for clinical assessment of those affected by adult participants with hemophilia.

Some of the tests (such as the Unipedal Stance Test or Four Square Step Test) have already been studied in children with hemophilia or in participants with other diseases. Since hemophilia is a disease with specific effects, the measuring instruments must also be researched in this participant group. There is still a research gap that the investigators would like to close with this study. For the study, the investigators selected tests that are already being used on adult participants with hemophilia and have had good experiences in practice. The tests are safe and can be carried out with little strain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Hemophilia Types A or B
* Adult people ≥ 18 years
* Patients on prophylactic factor or non-factor replacement treatment, or on demand factor replacement treatment.
* Able to walk for 20 meters independently, with or without walking aid
* Signed informed consent to participate in the study

Exclusion Criteria:

* Severe health conditions like severe cardiovascular, pulmonary, neurological or musculoskeletal diseases.
* Unable to perform the assessments due to disability or language problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline (Day 1) followed after a minimum break of 48 hours by Follow up (Day 2).
  SPPB comprises three components: Standing balance (open stand, half tandem stand and tandem stand), timed four meter usual paced walk, and timed test of five sit-to-stands from a standard chair. Each component is scored from 0 to 4, with maximum of 12and timed test of five sit-to-stands from a standard chair.
Four Square Step Test (FSST) | Baseline (Day 1) followed after a minimum break of 48 hours by Follow up (Day 2).
  The FSST is a performance-based outcome measure assessing dynamic balance. The test set up consists of four walking sticks of the same width in a cross formation. Participants step into each square in a clockwise sequence and back anticlockwise as fast as possible while not being allowed to hit the sticks.
Timed up and Go (TUG) | Baseline (Day 1) followed after a minimum break of 48 hours by Follow up (Day 2).
  The TUG is a performance-based outcome measure that assesses lower extremity function, mobility, and fall risk. In this test, the participant starts in a seated position, with his back against a standard height chair, without armrest. The participant gets up and walks in a comfortable pace for 10 feet (three meters), turns around and returns to a seated position in the chair. The time to perform the task is measured in seconds. Shorter time indicates better mobility.
Unipedal Stance Test (UST) | Baseline (Day 1) followed after a minimum break of 48 hours by Follow up (Day 2).
  The UST is a balance assessment that is widely used in clinical settings to monitor neurological and musculoskeletal conditions. Abnormal values may indicate conditions that may impair balance and will quantify balance status for those who are at increased risks for fall. The test is performed barefoot, hands crossed over the chest and once with eyes open and once with eyes closed. Patient stands on one leg unassisted; time begins when opposite foot leaves the ground. Time stops immediately when arms are uncrossed, the raised foot is used to maintain balance or touches the ground, weight-baring foot is moved, 45 second have elapsed or when eyes were opened on eyes closed trial. Each condition (eyes open or eyes closed) is performed three times, alternatively.
30-Second Stair Stand Test | Baseline (Day 1) followed after a minimum break of 48 hours by Follow up (Day 2).
  The 30-Second Chair Stand Test measures the muscle function of the lower extremity by counting how many times a patient rises from a seated position to a full stand at his/her own pace
1 kg Arm Lift Test | Baseline (Day 1) followed after a minimum break of 48 hours by Follow up (Day 2).
  The 1 kg arm lift test measures the muscle function of the upper extremity. It counts how many time a patient can lift a 1 kilogram weight above their head within 30 seconds at his/her own pace

SECONDARY OUTCOMES:
Short Form 36 | Baseline (Day 1)
  The Short Form 36 is a generic health related quality of life instrument consisting of 36 items pertaining to eight dimensions ('physical functioning', 'role physical functioning', 'bodily pain', 'general health perception', 'vitality', 'social functioning', 'role emotional functioning' and 'mental health'. The possible score ranges from 0 to 100 points, with 0 points representing the greatest possible health restriction, while 100 points indicate no health restriction.
  In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Hemophilia Activities List | Baseline (Day 1)
  The Hemophilia Activities List measures the impact of hemophilia on self-perceived functional abilities in adults. It contains 42 multiple choice questions in seven domains: Lying/sitting/kneeling/standing (8 items), Functions of the legs (9 items), Functions of the arms (4 items), Use of transportation (3 items), Self-care (5 items), Household tasks (6 items), Leisure activities and sports (7 items). The final version of the HAL has good internal consistency and convergent validity and gives the clinician insight into a patient's self-perceived ability to perform activities of daily life. The possible scores range from 0 to 100, where 0 represents the worst possible functional status and 100 the best possible functional status.
Hemophilia Joint Health Score Version 2.1 | Baseline (Day 1)
  The Hemophilia Joint Health Score2.1 includes swelling, duration (of swelling), muscle atrophy, crepitus on motion, flexion loss, extension loss, joint pain, strength, and global gait.
  For each of the Elbow, Knee and Ankle joints (left / rigth), the following items are scored: swelling (scored 0-3), duration of swelling (0-1), muscle atrophy (0-2), crepitus on motion (0-2), flexion loss (0-3), extension loss (0-3), joint pain (0-2), and strength (0-4). The maximum score for an individual index joint is 20. Gait is scored 0 to 4. The maximum HJHS total score is 124, with a higher score indicating worse joint health.

CONTACTS AND LOCATIONS:
Overall Officials: Ruud Knols, PhD, Principal Investigator — University of Zurich
Locations (1):
- Ruud Knols, Zurich, Switzerland